CLINICAL TRIAL: NCT05402436
Title: Breast Screening Atypia and Subsequent Development of Cancer: an Observational Analysis of the Sloane Database in England (Sloane Atypia Cohort Study)
Brief Title: Breast Screening Atypia and Subsequent Development of Cancer in England
Status: Completed | Type: Observational
Sponsor: University of Warwick (Other)
Collaborators: University Hospitals Coventry and Warwickshire NHS Trust (Other); King's College London (Other); The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Sian Taylor-Phillips, Professor of Population Health, University of Warwick
Other Study IDs: SOC.04/20-21
Record Dates: First submitted 2022-05-24; First posted 2022-06-02 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: Screening; Observational
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Women attending Breast Cancer Screening in England with an atypia diagnosis: Women attending Breast Cancer Screening in England with an atypia diagnosis between 1st January 2003 and 30th June 2018
  Interventions: Other: A diagnosis of atypia as part of the English screening programme

INTERVENTIONS:
Other: A diagnosis of atypia as part of the English screening programme — An atypia diagnosis of either ADH (including AIDEP), LISN (both ALH and LCIS) or FEA

SUMMARY:
During breast screening, atypical epithelial proliferations (atypia) can be detected. These are not cancer, but may mean that a woman is more likely to develop breast cancer in the future. This study explores how atypia develop into breast cancer in terms of number of women, time to cancer development, cancer type and severity, and whether this varies for different types of atypia. The results will be used to create new guidelines for how women with atypia should be followed up.

DETAILED DESCRIPTION:
In England, breast cancer screening is offered every three years to women aged 50 to 70. In an increasing number of women atypical epithelial proliferations (atypias) are detected. Atypias are a heterogeneous group of abnormalities, which are not cancer but carry a low but significant rate of associated malignancy. Detecting these lesions has uncertain benefit because of insufficient evidence on their risk of subsequent development into breast cancer. This information is key to optimising follow-up and subsequent screening. This study undertakes the first analysis of the Sloane atypia data by reporting the proportion of women with atypia who develop breast cancer by type of atypia (atypical ductal hyperplasia (ADH) or atypical intraductal epithelial proliferation (AIDEP), flat epithelial atypia (FEA), and lobular in situ neoplasia (LISN: atypical lobular hyperplasia (ALH) and lobular carcinoma in situ (LCIS)) and in what time frame.

This large-scale study of atypia uses the English screening programme data from the Sloane cohort study. The Sloane atypia project is a prospective cohort of atypia diagnosed through the UK NHS Breast Screening Programme from April 2003 to the present. For this analysis, English screening units are included with radiology, histopathology, surgery and radiotherapy proformas. Subsequent development of breast cancer has been identified by matching women by NHS number and date of birth to the English Cancer Registry held by the National Cancer Registration and Analysis Service (NCRAS). The atypia cases are also matched to the Mortality and Birth Information System to collect mortality data for censoring follow-up, and the Breast Screening Data Repository for information on invitation and attendance at subsequent screening mammography appointments.

Study objectives are:

1. To characterise atypia in terms of type, method of investigation and women's demographics;
2. To determine breast cancer risk over time by type of atypia;
3. To characterise the nature of subsequent cancers detected, and their prognostic features;
4. To communicate results to clinicians and women;
5. To recommend changes to the NHS Breast Screening Programme quality standards.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epithelial atypia (ADH (including AIDEP), LISN (both ALH and LCIS) and FEA) in the Sloane database between 1st January 2003 and 30th June 2018

Exclusion Criteria:

* bilateral primary cases
* the "best prognosis" atypia of the bilateral primaries
* atypia with co-existing DCIS
* pleomorphic LCIS (as these are managed akin to DCIS)
* unknown type of atypia
* cases not from England
* patients without follow-up until 31 December 2018

Ages: 47 Years to 73 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with atypia diagnosed during breast cancer screening in England between 1st January 2003 and 30th June 2018.
Sampling Method: Probability Sample
Enrollment: 3238 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Invasive breast cancer at 3 years following atypia diagnosis | Cumulative incidence of invasive breast cancer with all cause mortality as a competing risk at 3 years following atypia diagnosis
  Invasive breast cancer rate at 3 years following atypia diagnosis (representing the first round of screening) for all atypia, by type of atypia, by level of management off atypia, by three 5-year periods (deviding study period into 2003 to 2007, 2008 to 2012 and 2013 to 2018), by location (ipsilateral, contralateral), by age group, and by complete vs incomplete reporting of atypia cases by screening centres
Invasive breast cancer at 6 years following atypia diagnosis | Cumulative incidence of invasive breast cancer with all cause mortality as a competing risk at 6 years following atypia diagnosis
  Invasive breast cancer rate at 6 years following atypia diagnosis (representing the second round of screening) for all atypia, by type of atypia, by level of management off atypia, by three 5-year periods (deviding study period into 2003 to 2007, 2008 to 2012 and 2013 to 2018), by location (ipsilateral, contralateral), by age group, and by complete vs incomplete reporting of atypia cases by screening centres

SECONDARY OUTCOMES:
Invasive breast cancer at 1-year following atypia diagnosis | Cumulative incidence of invasive breast cancer with all cause mortality as a competing risk at 1-year following atypia diagnosis
  Invasive breast cancer rate at 1-year following atypia diagnosis (representing likely missed cancers at screening) for all atypia, by type of atypia, by level of management of atypia, by three 5-year periods (deviding study period into 2003 to 2007, 2008 to 2012 and 2013 to 2018), by location (ipsilateral, contralateral), by age group, and by complete vs incomplete reporting of atypia cases by screening centres
Invasive cancer or non-invasive cancer (Ductal carcinoma in situ (DCIS)) at 1 year following atypia diagnosis | Cumulative incidence of invasive breast cancer or DCIS with all cause mortality as a competing risk at 1 year following atypia diagnosis
  Rate of invasive breast cancer or DCIS at 1 year following atypia diagnosis for all atypia and by type and location of atypia
Invasive cancer or non-invasive cancer (Ductal carcinoma in situ (DCIS)) at 3 years following atypia diagnosis | Cumulative incidence of invasive breast cancer or DCIS with all cause mortality as a competing risk at 3 years following atypia diagnosis
  Rate of invasive breast cancer or DCIS at 3 years following atypia diagnosis for all atypia and by type and location of atypia
Invasive cancer or non-invasive cancer (Ductal carcinoma in situ (DCIS)) at 6 years following atypia diagnosis | Cumulative incidence of invasive breast cancer or DCIS with all cause mortality as a competing risk at 6 years following atypia diagnosis
  Rate of invasive breast cancer or DCIS at 6 years following atypia diagnosis for all atypia and by type and location of atypia

CONTACTS AND LOCATIONS:
Locations (1):
- Univesity of Warwick, Coventry, Warwickshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The investigators do not have Office for Data Release permissions to share these data more widely, but can assist other researchers in applying for access.

REFERENCES:
- [Background] Jenkinson D, Freeman K, Clements K, Hilton B, Dulson-Cox J, Kearins O, Stallard N, Wallis MG, Sharma N, Kirwan C, Pinder S, Provenzano E, Shaaban AM, Stobart H, McDonnell S, Thompson AM, Taylor-Phillips S. Breast screening atypia and subsequent development of cancer: protocol for an observational analysis of the Sloane database in England (Sloane atypia cohort study). BMJ Open. 2022 Jan 7;12(1):e058050. doi: 10.1136/bmjopen-2021-058050. PMID 34996804
- [Background] Freeman K, Mansbridge A, Stobart H, Clements K, Wallis MG, Pinder SE, Kearins O, Shaaban AM, Kirwan CC, Wilkinson LS, Webb S, O'Sullivan E, Jenkins J, Wright S, Taylor K, Bailey C, Holcombe C, Wyld L, Edwards K, Jenkinson DJ, Sharma N, Provenzano E, Hilton B, Stallard N, Thompson AM, Taylor-Phillips S. Evidence-informed recommendations on managing breast screening atypia: perspectives from an expert panel consensus meeting reviewing results from the Sloane atypia project. Br J Radiol. 2024 Feb 2;97(1154):324-330. doi: 10.1093/bjr/tqad053. PMID 38265306
- [Background] Freeman K, Jenkinson D, Clements K, Wallis MG, Pinder SE, Provenzano E, Stobart H, Stallard N, Kearins O, Sharma N, Shaaban A, Kirwan CC, Hilton B, Thompson AM, Taylor-Phillips S; Sloane Project Steering Group. Atypia detected during breast screening and subsequent development of cancer: observational analysis of the Sloane atypia prospective cohort in England. BMJ. 2024 Feb 1;384:e077039. doi: 10.1136/bmj-2023-077039. PMID 38302129